CLINICAL TRIAL: NCT06223061
Title: Global Evaluation of Cholecystectomy Knowledge and Outcomes
Acronym: GECKO
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: GlobalSurg 4 Edinburgh
Record Dates: First submitted 2023-11-30; First posted 2024-01-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Gallstone; Gallbladder Cancer; Bile Duct Injury
MeSH Terms: conditions — Gallstones; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cholecystectomy is amongst the most common surgical operations performed worldwide. Surgical candidates are treated for biliary pathologies, such as biliary colic, cholecystitis and gallstone pancreatitis. In patients who are deemed fit for surgery, cholecystectomy can be performed under three main settings: (1) emergency setting at index admission; (2) elective setting with no previous admissions; or (3) delayed setting with one or more previous gallbladder-related admissions.

The advent of laparoscopy fundamentally evolved biliary surgery and quickly became the "gold standard" approach. Recent multicentre collaborative studies have elucidated that the burden imposed on healthcare systems by laparoscopic cholecystectomies is primarily due to patient readmissions and complications arising from the operation, rather than perioperative mortality burden that was more commonly seen in open surgery. As a result, national and international societies have shifted their focus towards creating a culture of safety around this procedure, with the overarching goal of improving patient satisfaction and reducing hospital costs. The universal establishment of safe cholecystectomy is a complex process that relies not only on the operation itself, but also on various other factors such as promoting adequate training, improving hospital infrastructure, and enhancing perioperative patient care.

There remains a paucity of evidence around the variations of safe provision of laparoscopic surgery for gallbladder disease internationally, including low- and middle-income countries. To bridge this knowledge gap, the Global Evaluation of Cholecystectomy Knowledge and Outcomes (GECKO) study (GlobalSurg 4) will be an international collaborative effort, delivered by the GlobalSurg network, that will allow contemporaneous data collection on the quality of cholecystectomies using measures covering infrastructure, care processes and outcomes. It will be disseminated via contacts from the National Institute for Health and Care Research (NIHR) Global Surgery unit, leading emergency general surgeons and specialist organisations.

ELIGIBILITY:
Inclusion Criteria:

* Age: All adult patients (greater than or including 18 years of age).
* Procedure: Primary cholecystectomy, where this is the main procedure planned.
* Approach: Open, laparoscopic (standard and single-port), and robotic. Gasless laparoscopic and robotic approaches are inluded. Laparoscopic and robot converted cases are also eligible.
* Urgency: Elective, delayed and emergency procedures.

Exclusion Criteria:

* Procedure: Patients having a cholecystectomy as a part of another surgical procedure; for example, Whipple's procedure, bariatric, anti-reflux, or transplant operations, should be excluded.
* Indication: Patients with Mirizzi syndrome should be excluded.
* Return to theatre: Each patient should only be entered into the study once. Any patient returning to theatre and requiring a cholecystectomy for whatever indication, should not be included.
* Known gallbladder malignancy: when the diagnosis of gallbladder cancer is established pre-operatively, the patient should be excluded. However, if gallbladder cancer is found unexpectedly during or after cholecystectomy (i.e. on histology), the patient should be included.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, admitted to hospital within the pre-specified data collection periods, undergoing cholecystectomy as the index operation.
Sampling Method: Non-Probability Sample
Enrollment: 53708 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Compliance to pre-, intra-, and post-operative audit standards | 30-days from surgery
  Compliance to audit standards are defined as follows:
  1. Pre-operative: For patients with acute cholecystitis, surgeons may use the Tokyo Guidelines 18.
  2. Intraoperative: The use of the critical view of safety during laparoscopic cholecystectomy is the recommended approach to correctly identify relevant anatomy and minimize the risk of bile duct injuries
  3. Postoperative: 30-day readmission should be <10%.

SECONDARY OUTCOMES:
Quality of provision of cholecystectomy | 30-days of surgery
  The quality will be assessed according to the rates of overall complications defined as the presence of Grade I to grade V Clavien-Dindo complication.
Adverse events following cholecystectomy (e.g., bile duct injury) and their management. | 30-days of surgery
  Occurence of bile duct injury within 30-days of surgery will be defined according to the Strasberg Classification
Rates of unsuspected gallbladder cancer. | 1-year from surgery
  The rates of gallbladder cancer will be assessed at 1-year from the index surgery once the histology results are available.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] NIHR Global Health Research Unit on Global Surgery and the GlobalSurg Collaborative. Safety and equity in scaling minimally invasive surgery worldwide in 109 countries using cholecystectomy as a tracer procedure: a prospective cohort study. Lancet Glob Health. 2026 Feb;14(2):e199-e212. doi: 10.1016/S2214-109X(25)00476-0. PMID 41519150
- [Derived] Harrison E, Kathir Kamarajah S; NIHR Global Health Research Unit on Global Surgery. Global evaluation and outcomes of cholecystectomy: protocol for a multicentre, international, prospective cohort study (GlobalSurg 4). BMJ Open. 2024 Jul 25;14(7):e079599. doi: 10.1136/bmjopen-2023-079599. PMID 39059804